CLINICAL TRIAL: NCT03905603
Title: Relative Contributions of Predictors of Hyperandrogenism in Older vs. Young Women With PCOS
Acronym: SHK001
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Chris McCartney, Professor of Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21723
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Adrenocorticotropic Hormone; Cosyntropin; Ovidrel

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional physiological observational study.
Masking Description: No masking is involved in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACTH (Cosyntropin), rhCG (Ovidrel) (Experimental): ACTH (Cosyntropin) administered 250 mcg IV; rhCG (Ovidrel) administered 250 mcg IV
  Interventions: Drug: ACTH; Drug: rhCG

INTERVENTIONS:
Drug: ACTH — ACTH (Cosyntropin) 250 mcg will be given once during the study.
  Other Names: Cosyntropin
Drug: rhCG — rhCG (Ovidrel) 250 mcg will be given once during the study.
  Other Names: Ovidrel

SUMMARY:
The objective of the study is to determine the relative contributions of four established predictors of hyperandrogenism (luteinizing hormone [LH] secretion, ovarian response to recombinant human chorionic gonadotropin [r-hCG] administration, adrenal response to adrenocorticotropic hormone [ACTH] administration, and hyperinsulinemia) in older vs. young women with Polycystic Ovary Syndrome (PCOS) in a cross-sectional, physiological study. The investigators hypothesize that hyperinsulinemia is a stronger independent predictor of free testosterone (T) in older reproductive aged (vs. young) women with PCOS.

DETAILED DESCRIPTION:
PCOS is a highly prevalent reproductive disorder characterized by hyperandrogenism (HA) and oligo/anovulation. PCOS is also associated with metabolic syndrome, obesity and insulin resistance. In young women with PCOS, several factors contribute to HA: a) excess LH secretion, b) abnormal ovarian steroidogenesis, c) abnormal adrenal steroidogenesis, and d) hyperinsulinemia/ insulin resistance. Of interest, HA (and menstrual function) improves with age in PCOS. However, the relative contributions of the aforementioned HA-related factors in young adult vs. late reproductive-aged women with PCOS are not known. Identifying the most important predictor(s) of HA in older women with PCOS will be critically important for devising the most relevant therapeutic strategies for older women with PCOS. The investigators propose to determine the relative contributions of four established predictors of HA (LH secretion, ovarian response to r-hCG administration, adrenal response to ACTH administration, and hyperinsulinemia) in older vs. young women with PCOS in a physiological study. The investigators hypothesize that hyperinsulinemia is a stronger independent predictor of free testosterone (T) in older reproductive aged (vs. young) women with PCOS. In addition, the investigators hypothesize that, in older vs. young women with PCOS: a) ovarian response to r-hCG will be a weaker independent predictor of free T; b) mean LH will be a stronger independent predictor of free T; and c) the predictive ability of adrenal response to ACTH will be similar. This will be a cross-sectional physiological study. Ordinary Least Square (OLS) regression will be utilized to determine the relative contributions of 4 established predictors of HA in older vs. young women with PCOS. Statistical plans include intra-age group hypothesis testing, inter-age group hypothesis testing, and a ranking of the importance of predictors in each age group.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS aged 20-30 years and 40-49 years. Subject is considered to have PCOS if she has current or verifiable history of: a) clinical and/or biochemical evidence of hyperandrogenism plus b) oligomenorrhea (average menstrual cycle length >45 days or fewer than 9 menses/year) or irregular menstruation (substantially inconsistent menstrual cycle length). Note: For subjects aged 40-49 years, they will be allowed to participate if they have fewer than 10 menses/year (average menstrual cycle length >35 days) as long as they have a compelling past history of oligomenorrhea or irregular menstruation.
* Screening safety labs within normal reference ranges although mild abnormalities that are common in obesity and/or hyperandrogenism will not be grounds for exclusion (see exclusion criteria).
* Subjects must be willing and able to provide written informed consent.
* Willingness to strictly avoid pregnancy (using non-hormonal methods) during the time of the study
* Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

* Postmenopausal status (i.e., absence of periods for previous year plus elevated follicle stimulating hormone [FSH] level)
* Biochemical evidence for perimenopause as defined by an anti-Mullerian hormone <0.5 ng/mL. As an alternative, cycle day 3 FSH > 9 IU/L (with concomitant estradiol level >80 pg/mL), if this testing is available, will serve as evidence of perimenopause status. NOTE: If FSH >9 IU/L on screening (but it is not cycle day 3), FSH and estradiol will be repeated on cycle day 3.
* History of hysterectomy and/or bilateral oophorectomy
* BMI ≥ 40 kg/m2
* Inability to comprehend what will be done during the study or why it will be done.
* Being a study of older women with PCOS, children and men will be excluded.
* Pregnancy or lactation within the past 6 months. Subjects with a positive pregnancy test will be informed of the result by the screening physician.
* Prisoners.
* History of (or clinical evidence for) Cushing's syndrome or adrenal insufficiency.
* History of congenital adrenal hyperplasia or 17-hydroxyprogesterone (17-OHP) >200 ng/dL, which suggest the possibility of congenital adrenal hyperplasia. 17-OHP will be collected during follicular phase. NOTE: if a 17-OHP >200 ng/dL and is confirmed on repeat testing, an ACTH-stimulated 17-OHP <1000 ng/dL will be required for study participation.
* Total testosterone >150 ng/dL, which suggests the possibility of virilizing neoplasm.
* DHEA-S greater than 1.5 times the upper limit of normal range (mild elevations may be seen in PCOS, so elevations < 1.5 times the upper limit of normal will be accepted in these groups).
* Virilization
* Diagnosis of diabetes mellitus (DM), fasting glucose ≥ 126 mg/dL, or a hemoglobin A1c of ≥ 6.5%.
* Abnormal thyroid stimulating hormone (TSH). Subjects with stable and adequately-treated hypothyroidism, reflected by normal TSH values, will not be excluded.
* Moderate to severe hyperprolactinemia. Mild prolactin elevations may be seen in PCOS, and elevations < 1.5 times the upper limit of normal will be accepted in this group.
* Persistent liver abnormalities, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Mild transaminase elevations may be seen in women with obesity, so elevations <1.5 times the upper limit of normal will be accepted in this group.
* Hemoglobin level is less than 11 g/dL.
* Persistent hematocrit <36% and hemoglobin <12 g/dL.
* Subjects who remain anemic after two sequential months of ferrous gluconate (325 mg twice daily) will be excluded from study participation.
* Abnormal sodium, potassium, or bicarbonate concentrations or elevated creatinine concentration.
* Significant history of pulmonary dysfunction (e.g., asthma or COPD requiring intermittent systemic corticosteroid, pulmonary hypertension, etc.).
* History of known or suspected congestive heart failure.
* History of known or suspected ischemic heart disease or cerebrovascular disease.
* History of moderate to severe hypertriglyceridemia (triglyceride level > 500 mg/dL). Subjects with stable and adequately treated hypertriglyceridemia reflected by normal triglyceride values will not be excluded.
* History of breast, ovarian, or endometrial cancer.
* The cut off threshold for estimated dominant ovarian cyst size on the day of r-hCG injection will be 18 mm. Since the ultrasound will be assessed 3-4 days prior to r-hCG administration, we will estimate the size of the dominant follicle (at the time of r-hCG administration) using the typical rate of ovarian follicle growth of 1.4 mm per day. If the dominant follicle size exceeds the cut off threshold, the subject will be asked to repeat the transvaginal ultrasound: if menses begin within 3 weeks of the prior ultrasound, the ultrasound would be repeated during the new menstrual cycle. If menses do not occur within 3 weeks of the prior ultrasound, the ultrasound will then be scheduled at the subject's earliest convenience.
* Ovarian enlargement, defined by ovarian volume greater than 15 mm on transvaginal ultrasound. If the ovarian volume exceeds the cut off threshold, the participant will be given an option to repeat the transvaginal ultrasound in 2-3 months.
* History of venous thromboembolism (e.g. deep venous thrombosis (DVT), pulmonary embolism (PE)).
* History of blood clotting disorders (e.g., protein C, protein S, positive antiphospholipid antibodies).
* First-degree relative history of blood clotting disorder, unless the same disorder has been formally excluded for the study subject. Note: any abnormal labs may be repeated to exclude a lab error.
* No medications known to affect the reproductive system can be taken in the 2 months prior to screening and 3 months prior to the study. Such medications include oral contraceptive pills, metformin, progestins, glucocorticoids, anti-psychotics and/or mood stabilizers that are known to cause hormone abnormalities.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This is a study regarding PCOS, so only females will be eligible.
Enrollment: 144 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in calculated free testosterone concentrations | baseline, 30 mininutes and 1 hour after adrenocorticotropic hormone (ACTH), 24 hours after recombinant human chorionic gonadotropin (rhCG).
  pg/mL
Mean luteinizing hormone (LH) concentrations | overnight frequent blood sampling (every 10 mininutes for 12 hours)
  IU/L
Change in ovarian 17-hydroxyprogesterone to r-hCG | baseline, and 24 hours after receiving rhCG
  ng/mL
Change in adrenal 17-hydroxyprogesterone to ACTH | baseline, 30 minutes, and 60 minutes after ACTH
  ng/mL
Mean insulin level during oral glucose tolerance test | during 2 hours of oral glucose tolerance test
  uIU/mL

SECONDARY OUTCOMES:
Matsuda index | during 2 hours of glucose tolerance test
  It is an index calculated by using glucose and insulin levels
LH pulse frequency | overnight frequent blood sampling (every 10 minutes for 12 hours)
  pulses/hour
Change in dehydroepiandrosterone (DHEA) to r-hCG | baseline, and 24 hours after r-hCG
  ng/mL
Change in DHEA to ACTH | baseline, 30 minutes and 1 hour after ACTH
  ng/mL
Change in androstenedione to r-hCG | baseline, and 24 hours after r-hCG
  ng/mL
Change in androstenedione to ACTH | baseline, 30 minutes and 1 hour after ACTH
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Chris McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States